CLINICAL TRIAL: NCT02516683
Title: The Long Term Clinical Course of Postinfectious Irritable Bowel Syndrome After Shigellosis; A 10 Year Follow up Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 3-2011-0242
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Shigella Sonnei Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Shigella sonnei-exposed cohort: Shigella sonnei infection - A Shigella-exposed cohort of 124 hospital employees who had been infected by Shigella sonnei due to contaminated food in the employee-cafeteria in Gangnam Severance Hospital, Seoul, Korea, at December 2001.
  Interventions: Other: Shigella sonnei infection
- control cohort: A control cohort of age and sex-matched, non-infected 105 contemporary hospital employees.

INTERVENTIONS:
Other: Shigella sonnei infection — A Shigella-exposed cohort of 124 hospital employees who had been infected by Shigella sonnei due to contaminated food in the employee-cafeteria in Gangnam Severance Hospital, Seoul, Korea, at December 2001.
  Groups: Shigella sonnei-exposed cohort

SUMMARY:
Background: The incidence of postinfectious irritable bowel syndrome (PI-IBS) was reported to be in the range of 5-30%, but limited number of long-term follow-up results.

Objective: To investigate the long term clinical course of PI-IBS after Shigellosis.

Setting: A Shigellosis outbreak in a tertiary referral hospital with about 2,000 employees in Korea at 2001.

Patients: A Shigella-exposed cohort of 124 hospital employees who had been infected by Shigella sonnei due to contaminated food in the employee-cafeteria in Gangnam Severance Hospital, Seoul, Korea, at December 2001. A control cohort of age and sex-matched, non-infected 105 contemporary hospital employees.

Measurements: Questionnaire survey for bowel symptoms at 1, 3, 5, 8 and 10 years after outbreak.

DETAILED DESCRIPTION:
Postinfectious-IBS (PI-IBS) can be defined as the acute onset of new IBS symptoms in an individual, who has not previously met the criteria for IBS, immediately following an acute illness characterized by 2 or more of the following: fever, vomiting, diarrhea, or a positive bacterial stool culture.

Our group previously have reported clinical course of PI-IBS in a homogenous cohort which was comprised of patients recovered from Shigellosis. And in current study, we finally report a collective result of 10-year long-term follow-up of our small, but well-followed, homogenous cohort of PI-IBS after Shigellosis.

ELIGIBILITY:
Inclusion Criteria:

* Shigella sonnei infected patients

Exclusion Criteria:

* refused to participate in these surveys
* pregnant or had history of abdominal surgery or chronic organic gastrointestinal disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a Shigellosis outbreak took place at Gangnam Severance Hospital in Seoul, Korea, due to the consumption of contaminated food in the hospital cafeteria for employees. The causative pathogen was Shigella sonnei, and a total of 181 patients were diagnosed and treated for Shigellosis. After the termination of Shigellosis outbreak, we could establish a cohort of the Shigella-exposed group for serial surveys. The initially established Shigella-exposed cohort was comprised of 143 subjects, and we also could recruited the control group as age- and sex-matched healthy volunteers who were also hospital employees at same period and had not been infected, nor exposed to causal food.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2001-12; Primary Completion 2011-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Questionnaire survey for bowel symptoms | up to 10 years after outbreak

CONTACTS AND LOCATIONS:
Overall Officials: Young Hoon Youn, MD, PhD, Principal Investigator — Yonsei University